CLINICAL TRIAL: NCT05246800
Title: The Effectiveness of a Non-guided Mindfulness Application on Perceived Stress in a Non-clinical Dutch Population: a Randomized Controlled Trial
Brief Title: The Effectiveness of a Mindfulness Application on Perceived Stess
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Leonieke Kranenburg, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METC 2017-1117
Record Dates: First submitted 2022-01-31; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: mHealth; Mindfulness; Stress; Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT) was performed, comparing the experimental group that made use of a structured 8-week mHealth mindfulness program and a control group after 8 weeks, with follow-up after six months.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): a structured 8-week mHealth mindfulness program.
  Interventions: Other: Structured 8-week mHealth mindfulness program
- Control group (No Intervention): The control group was suggested to read the information about stress and burnout on the website of the TV-programme.

INTERVENTIONS:
Other: Structured 8-week mHealth mindfulness program — The mindfulness application was developed by Minddistrict The content of the app was developed by professionals in the field of mental healthcare and based on the principles of MBSR and MBCT The app consisted of a structured program, with chapters on psycho-education on mindfulness and the importance of practicing; acting on auto-pilot, conscious attention; non-judgmental attention, awareness; doing versus being-modus; attention for breath and body, conscious response; acceptance; a mindful attitude towards thoughts; applying mindfulness in daily life and staying mindful.
  Arms: Experimental group

SUMMARY:
Mindfulness has become increasingly popular and positive outcomes have been reported for mindfulness-based interventions (MBIs) in reducing stress. The aim of this study is to investigate if a non-guided mindfulness mobile phone application can decrease perceived stress in a non-clinical Dutch population over the course of eight weeks, with follow-up at six months.

DETAILED DESCRIPTION:
Background:

Mindfulness has become increasingly popular and positive outcomes have been reported for mindfulness-based interventions (MBIs) in reducing stress. These findings make room for innovative perspectives on how MBIs could be applied, for instance through mHealth.

Objectives:

The aim of this study is to investigate if a non-guided mindfulness mobile phone application can decrease perceived stress in a non-clinical Dutch population over the course of eight weeks, with follow-up at six months.

Methods:

A randomized controlled trial (RCT) was performed, comparing the experimental group that made use of a structured 8-week mHealth mindfulness program and a control group after 8 weeks, with follow-up after six months. Participants were recruited via a national television program. The primary outcome measure was perceived stress as measured by the Perceived Stress scale (PSS), secondary outcomes were symptoms of burnout (VAS) and psychological symptoms (measured by the four-dimensional symptom questionnaire ; 4DSQ at follow-up). Outcomes were analyzed using a multilevel regression model.

ELIGIBILITY:
Inclusion criteria:

>18 years

Exclusion criteria:

There were no other eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Change in perceived stress levels between baseline, end of program and after six months | baseline (before randomization), at the end of the program (eight weeks after randomization) and six months after randomization
  Measured with Perceived stress scale (PSS). The 14 item Dutch version was used. All items are rated on a 4-point Likert scale, with higher scores meaning more perceived stress.

SECONDARY OUTCOMES:
Change in burnout symptoms between baseline, end of program and after six months | baseline (before randomization), at the end of the program (eight weeks after randomization) and six months after randomization
  Measured with Visual analogue scale (VAS). Each symptom was rated on a 0-100 scale, with higher scores meaning higher difficulty.
Change in Four dimensional symptoms: : Distress (16 items), Depression (6 items), Anxiety (12 items) and Somatization between baseline, end of program and after six months | baseline (before randomization), at the end of the program (eight weeks after randomization) and six months after randomization
  Measured with Four dimensional symptom questionnaire (4DSQ). The 4DSQ consists of 50 items rated on a 4-point Likert scale. The 50 items can be grouped into four dimensions: Distress (16 items), Depression (6 items), Anxiety (12 items) and Somatization (16 items). Sum scores are calculated for each dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Leonieke Kranenburg, Principal Investigator — Department of Psychiatry, section Medical Psychology
Locations (1):
- Erasmus University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kranenburg LW, Gillis J, Mayer B, Hoogendijk WJG. The Effectiveness of a Nonguided Mindfulness App on Perceived Stress in a Nonclinical Dutch Population: Randomized Controlled Trial. JMIR Ment Health. 2022 Mar 18;9(3):e32123. doi: 10.2196/32123. PMID 35302504